CLINICAL TRIAL: NCT04862403
Title: The Effect of Umbilical Cord Clamping Distance on Cord Separation Time and Microbial Colonization: Randomized Controlled Study
Brief Title: The Effect of Umbilical Cord Clamping Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Deniz Akyıldız, Assistant professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Cord Clamping Distance
Record Dates: First submitted 2021-03-29; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Newborn; Infection; Umbilical Cord Infection
Keywords: colonization; midwives; newborn; separation time; umbilical cord
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group I (Experimental): In intervention group I - clamped at a distance of 2 cm - umbilical cord was measured 2 cm from the abdominal wall in the delivery room and clamped. This procedure was carried out by a single researcher using a 2 cm standard measuring tool (cut-to-size ruler) prepared before hand. In order to ensure standardization, this tool was cleaned with a disinfectant and used to measure the umbilical clamp distance of all newborns in the intervention group I.
  Interventions: Procedure: Umbilical cord clamping distance
- Intervention group II (Experimental): In intervention group II - clamped at a distance of 3 cm - umbilical cord was measured 3 cm from the abdominal wall in the delivery room and clamped. This procedure was carried out by a single researcher using a 3 cm standard measuring tool (cut-to-size ruler) prepared before hand. In order to ensure standardization, this tool was cleaned with a disinfectant and used to measure the umbilical clamp distance of all newborns in the intervention group II.
  Interventions: Procedure: Umbilical cord clamping distance
- Control group (No Intervention): Control group - clamped without measuring - no intervention was made in defining the distance at which the umbilical cord of the newborn would be clamped. Another healthcare workers measured the distance at which the umbilical cord had been clamped. The same researcher used a standard measuring tape to measure the distance between the umbilical cord to the clamping point.

INTERVENTIONS:
Procedure: Umbilical cord clamping distance — Intervention group I: Umbilical cord clamped at a distance of 2cm Intervention group II: Umbilical cord clamped at a distance of 3cm Control group: Usual care (clamped without measurement).
  Arms: Intervention group I; Intervention group II

SUMMARY:
A randomized control trial was conducted to test the effect of umbilical cord clamping distance on cord separation time and umbilical cord microbial colonization in neonates.

DETAILED DESCRIPTION:
Among the indicators of a country's level of development is the neonatal mortality rate. This rate reveals the extent of a country's economic development and how this affects health. One of the main causes of neonatal mortality is infection-related fatalities. Every year, approximately 700,000 neonatal deaths occur from bacterial infections.Navel cord infections comprise a large part of neonatal infections.

The umbilical cord is clamped and cut off at a distance of 2-3 cm from the newborn's abdominal wall after birth, after which its function is terminated. The necrotic tissue remaining in the newborn's umbilical cord provides an ideal environment for bacterial growth. The umbilical cord dries out and falls in the interval between postpartum 5-15 day. The prolongation of the umbilical cord falling time increases the possibility of developing bacterial infection. The umbilical cord microbial colonization was usually detected on 5th and 7th days after birth.

Since the time the umbilical cord falls off directly affects the health of the newborn, it is important to understand the factors that can affect this time. The literature reveals studies on umbilical cord separation times, most of which are devoted to comparing various techniques of caring for the cord. No study however has been discovered that has examined the effect of the distance between the abdominal wall of the newborn and the cord clamping site. It is believed that the clamping distance of the umbilical cord may be among the factors that have an impact on the separation time of the cord. Also, although midwives are responsible for the clamping and cutting of the umbilical cord, it is observed that there is no measuring instrument that is used in this procedure and the cord is clamped by eyeball estimation. There is no standard practice and there are also differences between the practices of midwives. This situation and the lack of adequate information in the literature on cord clamping distance pointed to the need for conducting a study in this context.

This study was intended to determine the effect of umbilical cord clamping distance on the cord separation time and on microbial colonization in the umbilical cord.

It was tested the hypotheses that there is no difference between the intervention and control groups of newborns after the umbilical cord clambing distance intervention, the cord separation time and on microbial colonization outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Being at 38-42 weeks of gestation, being 18 years of age and over, having primary school education, being able to speak and understand Turkish, having no communication problems, not having a history of active or previous vaginal infection, living in the metropolitan area of Kahramanmaras, accepting home visits during the research process, and agreeing to participate in the research.

Exclusion Criteria:

* Cesarean delivery, premature membrane rupture, newborns with severe congenital anomalies, severely ill infants requiring hospitalization immediately after birth, and babies born with a birth weight of less than 1500 g.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Umbilical cord separation time | 20th day after the birth
  assessed using the Umbilical Cord Follow-Up on Twentieth Day Form. This form consists of 17 questions prepared to investigate the umbilical cord separation time on the postpartum 20th day of the newborns in the intervention I, II, and control group. On the 20th day after birth, the mothers were called by mobile phone and information was obtained.
Umbilical cord microbial colonization | 7th day after the birth
  assessed with swab was taken from the umbilical cord on the 7th day. At home visits on the 7th postnatal day, a swab was taken from the umbilical cords of all newborns for microbial colonization. If the newborn's umbilical cord fell off on the 7th day postpartum visit, a swab was still taken. Umbilical swabs collected using transport swabs were transported to laboratory for culture. The result of the swab sample was taken 48 hours after the laboratory and it was determined whether there was colonization or not.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Akyıldız, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University; Ayden Çoban, Prof., Study Director — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lawn JE, Blencowe H, Oza S, You D, Lee AC, Waiswa P, Lalli M, Bhutta Z, Barros AJ, Christian P, Mathers C, Cousens SN; Lancet Every Newborn Study Group. Every Newborn: progress, priorities, and potential beyond survival. Lancet. 2014 Jul 12;384(9938):189-205. doi: 10.1016/S0140-6736(14)60496-7. Epub 2014 May 19. PMID 24853593
- [Background] Stewart D, Benitz W; COMMITTEE ON FETUS AND NEWBORN. Umbilical Cord Care in the Newborn Infant. Pediatrics. 2016 Sep;138(3):e20162149. doi: 10.1542/peds.2016-2149. PMID 27573092
- [Background] Duchowska A, Azsukowski P. Remarks on the length of umbilical arteries inhuman umbilical cord. A preliminary report. Archives of Perinatal Medicine. 2012;18(3):169-172.
- [Background] Ganatra HA, Zaidi AK. Neonatal infections in the developing world. Semin Perinatol. 2010 Dec;34(6):416-25. doi: 10.1053/j.semperi.2010.09.004. PMID 21094416
- [Background] Karumbi J, Mulaku M, Aluvaala J, English M, Opiyo N. Topical umbilical cord care for prevention of infection and neonatal mortality. Pediatr Infect Dis J. 2013 Jan;32(1):78-83. doi: 10.1097/INF.0b013e3182783dc3. PMID 23076382
- [Background] Arifeen SE, Mullany LC, Shah R, Mannan I, Rahman SM, Talukder MR, Begum N, Al-Kabir A, Darmstadt GL, Santosham M, Black RE, Baqui AH. The effect of cord cleansing with chlorhexidine on neonatal mortality in rural Bangladesh: a community-based, cluster-randomised trial. Lancet. 2012 Mar 17;379(9820):1022-8. doi: 10.1016/S0140-6736(11)61848-5. Epub 2012 Feb 8. PMID 22322124
- [Background] Abbaszadeh F, Hajizadeh Z, Jahangiri M. Comparing the Impact of Topical Application of Human Milk and Chlorhexidine on Cord Separation Time in Newborns. Pak J Med Sci. 2016 Jan-Feb;32(1):239-43. doi: 10.12669/pjms.321.8223. PMID 27022383
- [Derived] Akyildiz D, Coban A. How the Clamping Distance of the Umbilical Cord affects Microbial Colonization and Cord Separation Time: A Randomized Trial. P R Health Sci J. 2023 Mar;42(1):50-56. PMID 36941099